CLINICAL TRIAL: NCT07074158
Title: Identification of Microbial and Cytokine Signatures in Long COVID Patients: A Case-control Study of Long COVID Patients With Healthy Individuals
Brief Title: Microbial and Cytokine Signatures in Long COVID Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Palo Alto Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2024.133EXP
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will also be stored for future comparative studies of additional immune profiles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long COVID Subjects: Long COVID patients with a duration of illness longer than 6 months or longer will be included in the study.
- Healthy Controls: Healthy controls, matched by age to a long COVID subject (+/-10 years and preferably by sex).

SUMMARY:
We aim at identifying potential biomarkers in plasma indicative of post-acute coronavirus SARS-CoV-2 Syndrome (Long COVID). Our case-control study will compare Long COVID patients to healthy patients from Sutter Health.

DETAILED DESCRIPTION:
Two measures will be obtained from participants' plasma:

1. microbial signatures using Karius' agnostic metagenomic assay via microbial cell-free DNA (mcfDNA) sequencing (kariusdx.com)
2. cytokine signatures using 71-plex and 18-plex assays (evetechnologies.com).

The diagnostic utility of the potential biomarkers, including signatures derived from microbial cell-free DNA fragments found in plasma and plasma cytokines, will be evaluated independently and in various combinations to determine whether and to what extent we can accurately identify Long COVID patients. Moreover, we plan to leverage the Karius Test and the underlying Karius microbial cell-free DNA technology to determine whether there is evidence of more frequent reactivations of latent infections in patients with long COVID compared to matched healthy control. Plasma samples will also be stored for future comparative studies of additional immune profiles.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18-year-old
* English speaking (per Sutter medical records information)
* Ability and willingness to provide signed Consent Form
* Ability to comply with the study protocol
* Ability to attend the study visit, complete questionnaires, have blood collected and tested And, either Long-COVID or Healthy control as described below
* Long-COVID patient Cohort (n=75)

  * Sutter patient who is a patient from Sutter Health Holistic/Integrative Medicine clinic
  * Documentation of a long-COVID diagnosis (U09.9) for patient's initial visit in clinic between 01/01/2021 and 06/30/2024.
  * Presence of active and ongoing long-COVID symptoms
  * Ongoing long-COVID symptoms consistently present over the previous 6 months or longer
  * Presence of the following long-COVID symptoms (a, b, and c plus either d or e) affecting you more than 50% of your life:

    1. Fatigue that does not go away with rest.
    2. Post-exertional malaise ((worsening of your symptoms following cognitive, emotional, physical efforts)
    3. Unrefreshing sleep (sleep is not restorative)
    4. Brain "fog" (e.g., difficulty with finding words or mental tasks)
    5. Postural Orthostatic Hypotension (e.g., lightheadedness, dizziness, and/or palpitations with sitting up or standing up positions).
* Healthy controls with no Long COVID syndrome (n=75)

  * Sutter Health patients
  * Matched by age to a long COVID subject (+/-10 years and preferably by sex).

Exclusion Criteria:

* Pregnant or nursing woman
* Alcohol or another drug abuse ongoing within one year
* Severe depression or acute suicidal ideation
* Bipolar disorder, schizophrenia, or other psychosis
* History of malignancy, except basal cell carcinoma
* History of significant autoimmune disorder:

  * Addison disease
  * Dermatomyositis
  * Graves' disease
  * Multiple sclerosis
  * Myasthenia gravis
  * Pernicious anemia
  * Rheumatoid arthritis
  * Sjögren syndrome
  * Systemic lupus erythematosus
  * Type I diabetes
  * Celiac disease
* Active pulmonary infection (active pneumonia)
* Chronic kidney disease
* Chronic liver disease
* Chronic lung disease
* Pulmonary fibrosis
* Interstitial pneumonitis
* Uncontrolled asthma
* Chronic obstructive pulmonary disease (COPD)
* Reactive arthritis
* Immunocompromised conditions or weaken immune system:

  * Cancer under treatment or treated within one year of enrollment
  * AIDS
  * Transplant patient
* Biologicals impacting the immune system
* Taking immunosuppressor
* Neurologic conditions:

  * Dementia or other neurological conditions
  * Acute Spinal Cord Injury
  * Alzheimer's Disease
  * Amyotrophic Lateral Sclerosis (ALS)
  * Ataxia
  * Cerebral Aneurysm diagnosed within one year of enrollment
  * Epilepsy and Seizures uncontrolled with medication
* Heart conditions:

  * Congestive heart failure
  * Myocardial infarction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will focus on participants with a diagnosis code for long-COVID (U09.9) in their Sutter EMR and healthy controls who are Sutter Health's patients.
  It will enroll 75 patients diagnosed with long-COVID and 75 matched healthy controls respectively.
  Healthy controls will be matched 1:1 to long-COVID patients for age (+/-10 years and preferably by sex).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2026-07-13 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Metagenomics | Baseline
  In this proof-of-concept study, we want to test the hypothesis that mcfDNA has diagnostic utility as a biomarker for long COVID patients by applying the agnostic metagenomic sequencing approach.
Cytokines | Baseline
  Cytokine signatures have been associated with disease severity in patients with chronic fatigue syndrome (Montoya et al, Proc Natl Acad Sci U S A. 2017 Aug 22;114(34): E7150-E7158.). We want to test the hypothesis that cytokine profiles may serve as surrogate biomarkers for Long COVID.
Metadata analysis | Baseline
  Analysis of microbial-cell-free DNA and cytokine to identity meta-signatures associated with Long COVID and/or Long COVID severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Montoya, Principal Investigator — Sutter Health, Palo Alto Medical Foundation
Locations (1):
- Sutter Health Palo Alto Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No